CLINICAL TRIAL: NCT01286207
Title: Long-Term Exposure to Rizatriptan 5-mg and 10-mg Oral Tablet (Combined Protocols 022, 025, 029)
Brief Title: Long-Term Exposure to Rizatriptan 5-mg and 10-mg Oral Tablet (Combined Extension Protocols MK-0462-022, MK-0462-025, MK-0462-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0462 Pooled 022/025/029
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Migraine Disorders
Keywords: Migraine headache
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rizatriptan 5 mg (Experimental): Rizatriptan 5 mg orally once for treatment of index migraine attack, followed by two additional doses within 24 hours of the initial dose for migraine recurrence(s)
  Interventions: Drug: Rizatriptan 5 mg
- Rizatriptan 10 mg (Experimental): Rizatriptan 10 mg orally once for treatment of index migraine attack, followed by two additional doses within 24 hours of the initial dose for migraine recurrence(s)
  Interventions: Drug: Rizatriptan 10 mg
- Standard Care (Active Comparator): Standard care at onset of migraine attack
  Interventions: Drug: Standard Care

INTERVENTIONS:
Drug: Rizatriptan 5 mg — Rizatriptan 5 mg orally once for treatment of index migraine attack, followed by two additional doses within 24 hours of the initial dose for migraine recurrence(s)
  Other Names: MK-0462, Maxalt
  Arms: Rizatriptan 5 mg
Drug: Rizatriptan 10 mg — Rizatriptan 10 mg orally once for treatment of index migraine attack, followed by two additional doses within 24 hours of the initial dose for migraine recurrence(s)
  Other Names: MK-0462, Maxalt
  Arms: Rizatriptan 10 mg
Drug: Standard Care — Active standard care
  Arms: Standard Care

SUMMARY:
This record describes pooled data for three extension studies: MK-0462-022 (NCT00897949); MK-0462-025 (NCT00899379); and MK-0462-029 (NCT00897104). These studies examined the long-term safety and efficacy of rizatriptan used for the treatment of acute migraine and migraine recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Participant took part in study MK-0462-022, MK-0462-025, or MK-0462-029
* History of migraine headache

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1959 (Actual)
Dates: Start 1995-03; Primary Completion 1997-05 (Actual); Study Completion 1997-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants that completed protocol MK-0462-022 (NCT00897949), MK-0462-025 (NCT00899379), or MK-0462-029 (NCT00897104) and consented to continue in the studies up to 12 months were included in this pooled extension data.
Period: Overall Study
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Started | 751 | 857 | 351
Completed | 453 | 609 | 261
Not Completed | 298 | 248 | 90
Not completed — Adverse Event | 27 | 41 | 8
Not completed — Lost to Follow-up | 49 | 43 | 20
Not completed — Withdrawal by Subject | 93 | 79 | 41
Not completed — Lack of Response | 92 | 38 | 8
Not completed — Other | 37 | 47 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care | Total
Number analyzed (Participants) | 751 | 857 | 351 | 1959
Age, Continuous [Mean (Full Range); unit: years] | 41.6 [18 to 66] | 41.1 [18 to 65] | 40.7 [18 to 64] | 41.2 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 643 | 727 | 300 | 1670
  Male | 108 | 130 | 51 | 289

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patient's Headaches With Pain Relief at 2 Hours After the Initial Dose of Test Drug
Description: Headache severity was rated on a 4-point scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain) immediately before initial dose and at 2 hours thereafter. Pain relief was defined as a reduction of headache severity from grades 2/3 at baseline to 0/1.
Time Frame: 2 hours after initial dose of test drug
Population: All patients who took study medication and filled out their diary cards were included in the analysis of efficacy. No data were imputed.
Measure: Median (Inter-Quartile Range); unit: percent of headaches
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Number analyzed (Participants) | 606 | 815 | 325
percent of headaches | 80 [55.6 to 93.8] | 89.5 [75.0 to 98.0] | 69.6 [46.2 to 92.0]

2. Primary Outcome: Number of Participants With Serious Clinical Adverse Experiences
Description: Serious clinical adverse experiences (CAEs) are any adverse events (AEs) occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose.
Time Frame: Up to 12 months
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Number analyzed (Participants) | 711 | 834 | 334
participants
  With Serious CAEs | 13 | 17 | 10
  Without Serious CAEs | 698 | 817 | 324

3. Primary Outcome: Number of Participants With Drug-related Clinical Adverse Experiences
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs.
Time Frame: Up to 12 months
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Number analyzed (Participants) | 711 | 834 | 334
participants
  With drug-related CAEs | 288 | 456 | 139
  Without drug-related CAEs | 423 | 378 | 195

4. Primary Outcome: Number of Participants Who Discontinued Due to Clinical Adverse Experiences
Time Frame: Up to 12 months
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Number analyzed (Participants) | 711 | 834 | 334
participants
  Discontinued due to CAEs | 26 | 37 | 7
  Not discontinued due to CAEs | 685 | 797 | 327

5. Primary Outcome: Number of Participants With Drug-related Lab Adverse Experiences
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) laboratory adverse experience (LAE).
  A LAE is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
Time Frame: Up to 12 weeks
Population: All patients who took study medication and had lab test(s)were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Number analyzed (Participants) | 709 | 827 | 333
participants | 15 | 23 | 4

ADVERSE EVENTS:
Description: The 'total # participants affected' w/ Other AEs DOES include subjects w/ any AE (including SAEs) >1 event. The true overall # of subjects affected w/ only any NonSerious AE >5% is less than the # reported, but unable to be determined for this pooled extension period.
  Specific Other AEs reported DO NOT include SAEs and DO NOT include events <5%
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Standard Care
Serious Adverse Events (participants affected / at risk) | 13/711 | 17/834 | 10/334
Other Adverse Events (participants affected / at risk) | 492/711 | 679/834 | 267/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=711) | Rizatriptan 10 mg (N=834) | Standard Care (N=334)
Hernia, inguinal (General disorders) | 0 | 0 | 1 — Body as a whole/site unspecific (SOC)
Melanoma (General disorders) | 1 | 0 | 0 — Body as a whole/site unspecific (SOC)
Pain, abdominal (General disorders) | 0 | 1 | 2 — Body as a whole/site unspecific (SOC)
Pain, chest (General disorders) | 0 | 1 | 0 — Body as a whole/site unspecific (SOC)
Septicimea (General disorders) | 0 | 0 | 1 — Body as a whole/site unspecific (SOC)
Surgery, abdominal (General disorders) | 0 | 0 | 1 — Body as a whole/site unspecific (SOC)
Trauma (General disorders) | 1 | 0 | 0 — Body as a whole/site unspecific (SOC)
Embolism/infarction, pulmonary (Cardiac disorders) | 0 | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Gastrointestinal disorders) | 0 | 1 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, anal/rectal (Gastrointestinal disorders) | 0 | 1 | 0
Rectocele (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Neoplasm, thyroid, malignant (Endocrine disorders) | 1 | 0 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaphylaxis (Metabolism and nutrition disorders) | 0 | 1 | 0 — Metabolic/Nutritional/Immune (SOC)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 — Metabolic/Nutritional/Immune (SOC)
Fracture, elbow, right (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fracture, hip, right (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain, back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain, knee (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain, neck (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Trauma, cartilage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anxiety (Nervous system disorders) | 1 | 0 | 0 — Nervous System and Psychiatric (SOC)
Depression (Nervous system disorders) | 1 | 0 | 1 — Nervous System and Psychiatric (SOC)
Headache (Nervous system disorders) | 0 | 1 | 0 — Nervous System and Psychiatric (SOC)
Meningitis (Nervous system disorders) | 0 | 0 | 1 — Nervous System and Psychiatric (SOC)
Migraine (Nervous system disorders) | 1 | 3 | 3 — Nervous System and Psychiatric (SOC)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Neoplasm, skin, malignant (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Abortion (Reproductive system and breast disorders) | 0 | 1 | 0 — Urogenital System (SOC)
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 — Urogenital System (SOC)
Hypertrophy, uterine (Reproductive system and breast disorders) | 0 | 1 | 0 — Urogenital System (SOC)
Neoplasm, breast, malignant (Reproductive system and breast disorders) | 1 | 0 | 0 — Urogenital System (SOC)
Neoplasm, uterine, benign (Reproductive system and breast disorders) | 1 | 0 | 0 — Urogenital System (SOC)
Pregnancy (Reproductive system and breast disorders) | 0 | 1 | 0 — Urogenital System (SOC)
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 — Urogenital System (SOC)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=711) | Rizatriptan 10 mg (N=834) | Standard Care (N=334)
Asthenia/fatigue (General disorders) | 70 | 111 | 44 — Body as a Whole/Site Unspecific (SOC)
Pain, abdominal (General disorders) | 24 | 27 | 18 — Body as a Whole/Site Unspecific (SOC)
Pain, chest (General disorders) | 34 | 61 | 28 — Body as a Whole/Site Unspecific (SOC)
Diarrhea (Gastrointestinal disorders) | 21 | 32 | 18
Nausea (Gastrointestinal disorders) | 117 | 178 | 86
Vomiting (Gastrointestinal disorders) | 51 | 72 | 29
Pain, back (Musculoskeletal and connective tissue disorders) | 30 | 48 | 18
Dizziness (Nervous system disorders) | 69 | 135 | 35 — Nervous System and Psychiatric (SOC)
Headache (Nervous system disorders) | 62 | 100 | 42 — Nervous System and Psychiatric (SOC)
Insomnia (Nervous system disorders) | 21 | 31 | 17 — Nervous System and Psychiatric (SOC)
Paresthesia (Nervous system disorders) | 34 | 63 | 24 — Nervous System and Psychiatric (SOC)
Somnolence (Nervous system disorders) | 50 | 127 | 30 — Nervous System and Psychiatric (SOC)
Infection, respiratory, upper (Respiratory, thoracic and mediastinal disorders) | 78 | 114 | 46
Influenza (Respiratory, thoracic and mediastinal disorders) | 46 | 52 | 25
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 21 | 47 | 22
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 37 | 72 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.